CLINICAL TRIAL: NCT01697189
Title: An Educational Intervention to Promote Safe and Economic Truck Driving
Brief Title: An Educational Intervention to Promote Safe Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute of Occupational Health (Other)
Collaborators: University of Jyvaskyla (Other); Tampere University of Technology (Other); Taipale Telematics Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EISD-109378-FWF; EISD-109378-FWEF (Other Grant/Funding Number: Finnish Work Environment Fund)
Record Dates: First submitted 2010-11-05; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Driver Sleepiness
Keywords: professional drivers; sleepiness; stress; safe driving; training
MeSH Terms: conditions — Sleepiness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fatigue management training (Experimental): Experimental group subjects participated in a single half-day fatigue management training session.
  Interventions: Behavioral: Fatigue management training
- No fatigue management training (No Intervention): The control group subjects did not participate in the fatigue management training.

INTERVENTIONS:
Behavioral: Fatigue management training — Experimental group took part in a single half-day (4 hours) fatigue management training grounded on Problem Based Learning (PBL).
  Arms: Fatigue management training

SUMMARY:
The general aim of the study is to promote safe, economic, and environmental-friendly driving among long-haul truck drivers. To do this, the investigators will conduct an on-road study on i) the relationship of driver sleepiness and stress with driving behaviour and fuel consumption and ii) effectiveness of an educational intervention in mitigating sleepiness at the wheel. The educational intervention is designed to be employed by occupational health care professionals in the future. This solution clearly facilitates the implementation of the intervention into practice if it turns out to be effective.

The investigators specified research questions are the following:

* Do truck driver sleepiness and stress at the wheel reach levels that affect driving behaviour, fuel consumption and carbon emissions?
* What are the sources of sub-optimal arousal at the wheel in truck drivers?
* Can truck driver sleepiness be mitigated by an educational intervention, and if yes, does it improve driving behaviour and decrease fuel consumption and carbon emissions as well?

ELIGIBILITY:
Inclusion Criteria:

* working as a truck driver at the moment of the study
* having both day and night trips
* having at least 2 years of experience in truck driving

Exclusion Criteria:

* not fluent in Finnish (the intervention is in Finnish)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
driver sleepiness | one year
  Self-reported sleepiness measured by the the Karolinska Sleepiness Scale Questionnaire and behavioral sleepiness measured by the Observer Rating of Drowsiness (based on video materia).

SECONDARY OUTCOMES:
driver stress | one year
  Self-rating scale of stress and heart rate measures of stress (heart rate variability)
sleep | one year
  wrist-worn actigraphy and sleep diary based measures of sleep quantity, timing and quality
driving behaviour | one year
  vehicle movement-based measures of driving behaviour (speed, accelerations, deceleration)

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Sallinen, PhD, Principal Investigator — Finnish Institute of Occupational Health
Locations (1):
- Finnish Institute of Occupational Health, Helsinki, Finland